CLINICAL TRIAL: NCT01567904
Title: An Open-label, Pharmacokinetic, Pharmacodynamic, and Tolerability Study of AVE5026 Administered at Weight-adjusted Doses to Patients Less Than 18 Years of Age With a Central Venous Line (CVL)
Brief Title: Study of AVE5026 at Weight-adjusted Doses in Children With a Central Venous Line
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Decision from Sanofi to withdraw on a worldwide basis the Marketing Authorisation Applications for Semuloparin sodium in the adult indication
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PKM11204; 2011-005155-14 (EudraCT Number); U1111-1115-8281 (Other: UTN)
Record Dates: First submitted 2012-03-28; First posted 2012-03-30 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Thrombosis Prophylaxis (Risk of Thrombosis Due to Central Venous Line (CVL)
Keywords: thrombosis; Central Venous Line; CVL
MeSH Terms: conditions — Thrombosis | interventions — AVE 5026

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Age group from 12 to 18 (<) years (Experimental): Semuloparin sodium, weight-adjusted dose once daily for 6-30 days
  Interventions: Drug: Semuloparin sodium
- Age group from 6 to 12 (<) years (Experimental): Semuloparin sodium, weight-adjusted dose once daily for 6-30 days
  Interventions: Drug: Semuloparin sodium
- Age group from 2 to 6 (<) years (Experimental): Semuloparin sodium, weight-adjusted dose once daily for 6-30 days
  Interventions: Drug: Semuloparin sodium
- Age group from 3 months to 2 (<) years (Experimental): Semuloparin sodium, weight-adjusted dose once daily for 6-30 days
  Interventions: Drug: Semuloparin sodium
- Age group from birth to 3 (<) months (Experimental): Semuloparin sodium, weight-adjusted dose once daily for 6-30 days
  Interventions: Drug: Semuloparin sodium

INTERVENTIONS:
Drug: Semuloparin sodium — Solution for injection in single dose vials (10 mg/mL and 20 mg/mL)
  Subcutaneous injection
  Other Names: AVE5026

SUMMARY:
Primary Objective:

- To assess the pharmacokinetic (PK) and pharmacodynamic (PD) parameters of Semuloparin [AVE5026] (assessed from the anti-Xa activity of Semuloparin) in children in order to determine the dose to be assessed in a clinical efficacy/safety study in this population.

Secondary Objective:

- To assess the tolerability of Semuloparin when administered at a weight-adjusted, once daily dose for up to 30 days in patients less than 18 years of age with central venous line.

DETAILED DESCRIPTION:
The maximum study duration for a participant was 68 days broken down as follows:

* Screening period: up to 6 days,
* Treatment period: minimum 6 days and maximum 30 days,
* Follow-up period with an end of study visit performed 4 weeks (30 +/-2 days) post treatment.

Enrollment staggered by age group starting with the older children (≥12 years). In each younger age group, enrolment was planned to initiate only following a review by the Data Monitoring Committee (DMC) of the clinical safety data and available PK and PD data from the first 3 out of 7 children from the previous older age group. Enrollment of infants <3 months was planned to initiate after recruitment of all patients ≥3 months had been completed and all data analyzed by the DMC.

ELIGIBILITY:
Inclusion criteria :

* age between ≥38 gestational weeks and <18 years;
* Central Venous Line implanted for an expected duration ≥6 days from study enrolment;
* Patient hospitalized or able to receive daily injection for at least 6 days and provide plasma samples at Day 4, 5 and 6 at the pre-specified time points;
* Written informed consent signed by legal representative(s) in accordance with local regulation, and possibly assent form by the child (country/age specific).

Exclusion criteria:

* Patient for whom anticoagulant therapy was contraindicated;
* Planned treatment with other antithrombotic agents within 2 weeks prior to enrolment and during the course of the study;
* Any previous exposure to Semuloparin (e.g. previous enrolment in the current study);
* Documented history of heparin-induced thrombocytopenia;
* Severe thrombocytopenia (platelets <50 x 109/L);
* Active bleeding;
* Recent (less than 3 weeks prior to enrollment ) brain, spinal or ophthalmologic surgery;
* Uncontrolled hypertension characterized by a sustained systolic pressure or diastolic pressure greater than 2 standard deviations above the age-related norm;
* Severe hepatic disease (e.i. more than 2.5 times the upper limit for age of hepatic enzymes);
* Severe renal insufficiency (estimated creatinine clearance <30 ml/min using the Schwartz formula);
* Any condition that, in the opinion of the Investigator, would have exposed the patient to an unfavorable risk/benefit ratio;
* Presence or history of drug hypersensitivity;
* Any patient currently involved in another clinical trial with an investigational drug according to applicable regulations;
* Any patient or parent(s)/legal guardian(s) who, in the judgment of the Investigator, was likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development;
* Any patient or parent(s)/legal guardian(s) who could not be contacted in case of emergency;
* Pregnant or breast-feeding female;
* Female of childbearing potential who were unwilling to abstain from sexual intercourse and therefore were at risk of becoming pregnant and were not protected by highly effective contraceptive method of birth control and/or who were unwilling or unable to be tested for pregnancy.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Plasma concentrations of Semuloparin | 6 samples; 0.5-1h and 6h after D4 injection, 1.5-4h and 12h after D5 injection, just before and 8h after D6 injection
  A validated anti-Xa chromogenic enzyme assay, with addition of AT-III in excess was to be used to assess plasma concentrations of semuloparin.
  A full population PK model of semuloparin in children (including covariates assessment) was to be established and individual pharmacokinetic parameters were be estimated.
Pharmacodynamic activity (anti-Xa activity) of Semuloparin | 6 samples; 0.5-1h and 6h after D4 injection, 1.5-4h and 12h after D5 injection, just before and 8h after D6 injection
  A validated anti-Xa chromogenic enzyme assay, without addition of AT-III in excess, was to be used to assess pharmacodynamic activity (factor Xa inhibition) of semuloparin.
  A full population PK/PD model of semuloparin in children (including covariates assessment) was to be established and individual pharmacodynamic parameters were to be estimated.

SECONDARY OUTCOMES:
Safety parameters including bleeding | up to 30+/- 2 days post treatment
Safety parameters including transfusions requirement | up to 30+/- 2 days post treatment
Safety parameters including hemoglobin, platelet count | up to 30+/- 2 days post treatment
Safety parameters including liver and renal laboratory data | up to 30+/- 2 days post treatment
Safety parameters including serious adverse events | up to 30+/- 2 days post treatment
Safety parameters including non-serious adverse events | up to 30+/- 2 days post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 348001, Budapest, Hungary